CLINICAL TRIAL: NCT02044172
Title: The ProtecT Trial - Evaluating the Effectiveness of Treatments for Clinically Localised Prostate Cancer
Brief Title: Prostate Testing for Cancer and Treatment
Acronym: ProtecT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: University of Bristol (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HTA96/20/99; 20141297 (Registry Identifier: ISRCTN); NCT00632983 (obsolete NCT alias)
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Treatment; Screening; Surgery; Radiotherapy; Active monitoring
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Radical prostatectomy (Active Comparator): Radical prostatectomy
  Interventions: Procedure: Radical prostatectomy
- Conformal radiation therapy (Active Comparator): Conformal radiation therapy External beam radiation therapy
  Interventions: Radiation: Conformal radiation therapy
- Active monitoring (Active Comparator): Active monitoring of prostate specific antigen levels and disease surveillance
  Interventions: Other: Active monitoring

INTERVENTIONS:
Procedure: Radical prostatectomy — radical prostatectomy
  Arms: Radical prostatectomy
Radiation: Conformal radiation therapy — Conformal radiation therapy, external beam
  Arms: Conformal radiation therapy
Other: Active monitoring — Active monitoring of Prostate specific antigen levels and disease surveillance
  Arms: Active monitoring

SUMMARY:
RATIONALE: Radical prostatectomy is surgery to remove the entire prostate. Radiation therapy uses high-energy x-rays or other types of radiation to kill tumor cells. Sometimes the tumor may not need treatment until it progresses. In this case, active surveillance may be sufficient. It is not yet known which treatment regimen is more effective for localized prostate cancer.

PURPOSE: This randomized phase III trial is studying active monitoring to see how well it works compared with radical prostatectomy or radiation therapy in treating patients with localized prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess survival of patients with localized prostate cancer at 10 years and 15 years after treatment.
* To investigate disease progression (i.e., biochemical and clinical), treatment complications, and lower urinary tract symptoms in these patients.
* To investigate the psychosocial impact of cancer detection and treatment on these patients, including generic health status, quality of life, and sexual function.
* To estimate the resource use and costs of detection, treatment, and follow-up.
* To compare costs and outcomes of treatment in terms of survival and health-related quality of life.
* To collect samples suitable for basic science research (ProMPT study).

OUTLINE: This is a multicenter study. Patients are stratified by age (50-55 vs 56-59 vs 60-65 vs 66-69 years), Gleason score (6, 7, 8-10), and average result of recruitment and first biopsy prostate-specific antigen (PSA) tests (< 6 vs 6-9.9 vs ≥ 10 ng/mL). Patients are randomized or select a treatment to be followed up in a cohort study.

ELIGIBILITY:
Inclusion Criteria:

Fit for the treatments and estimates life expectancy of 10 years Registration with eligible primary care practice

Exclusion Criteria:

Unable to give written informed consent. Concomitant or past malignancy.

Ages: 50 Years to 69 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82849 (Actual)
Dates: Start 2001-06-01 (Actual); Primary Completion 2020-11-14 (Actual); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Disease specific mortality | Median 15 years follow up

SECONDARY OUTCOMES:
Overall survival | Median 15 years
Disease progression | Median 15 years
  Metastases
Treatment complications | Median 15 years
General health status | Median 15 years
Psychological state | Median 15 years
Symptoms | Median 15 years
Sexual function | Median 15years

CONTACTS AND LOCATIONS:
Overall Officials: Freddie C Hamdy, Principal Investigator — University of Oxford
Locations (8):
- United Kingdom (8):
  - Queen Elizabeth Hospital, Birmingham
  - Southmead Hospital, Bristol
  - Addenbrokes' Hospital, Cambridge
  - University Hospital of Wales, Cardiff
  - Western General Hospital, Edinburgh
  - Leicester General Hospital, Leicester
  - Freeman Hospital, Newcastle
  - Royal Hallamshire Hospital, Sheffield

REFERENCES:
- [Background] Lane JA, Hamdy FC, Martin RM, Turner EL, Neal DE, Donovan JL. Latest results from the UK trials evaluating prostate cancer screening and treatment: the CAP and ProtecT studies. Eur J Cancer. 2010 Nov;46(17):3095-101. doi: 10.1016/j.ejca.2010.09.016. PMID 21047592
- [Derived] Sushentsev N, Warren AY, Colling R, Verrill C, Pazukhina E, Blyuss O, Seibert TM, Barrett T, Mills IG, Bryant RJ, Donovan JL, Neal DE, Hamdy FC. Active Monitoring, Surgery, and Radiotherapy for Cribriform-Positive and Cribriform-Negative Prostate Cancer: A Secondary Analysis of the PROTECT Randomized Clinical Trial. JAMA Oncol. 2025 Dec 1;11(12):1512-1517. doi: 10.1001/jamaoncol.2025.4125. PMID 41100113
- [Derived] Donovan JL, Hamdy FC, Lane JA, Young GJ, Metcalfe C, Walsh EI, Davis M, Steuart-Feilding T, Blazeby JM, Avery KNL, Martin RM, Bollina P, Doble A, Doherty A, Gillatt D, Gnanapragasam V, Hughes O, Kockelbergh R, Kynaston H, Paul A, Paez E, Powell P, Rosario DJ, Rowe E, Mason M, Catto JWF, Peters TJ, Wade J, Turner EL, Williams NJ, Oxley J, Staffurth J, Bryant RJ, Neal DE. Patient-Reported Outcomes 12 Years after Localized Prostate Cancer Treatment. NEJM Evid. 2023 Apr;2(4):EVIDoa2300018. doi: 10.1056/EVIDoa2300018. Epub 2023 Mar 11. PMID 38320051
- [Derived] Hamdy FC, Donovan JL, Lane JA, Metcalfe C, Davis M, Turner EL, Martin RM, Young GJ, Walsh EI, Bryant RJ, Bollina P, Doble A, Doherty A, Gillatt D, Gnanapragasam V, Hughes O, Kockelbergh R, Kynaston H, Paul A, Paez E, Powell P, Rosario DJ, Rowe E, Mason M, Catto JWF, Peters TJ, Oxley J, Williams NJ, Staffurth J, Neal DE; ProtecT Study Group. Fifteen-Year Outcomes after Monitoring, Surgery, or Radiotherapy for Prostate Cancer. N Engl J Med. 2023 Apr 27;388(17):1547-1558. doi: 10.1056/NEJMoa2214122. Epub 2023 Mar 11. PMID 36912538
- [Derived] Sanghera S, Mohiuddin S, Coast J, Garfield K, Noble S, Metcalfe C, Lane JA, Turner EL, Neal D, Hamdy FC, Martin RM, Donovan JL; ProtecT study group. Modelling the lifetime cost-effectiveness of radical prostatectomy, radiotherapy and active monitoring for men with clinically localised prostate cancer from median 10-year outcomes in the ProtecT randomised trial. BMC Cancer. 2020 Oct 7;20(1):971. doi: 10.1186/s12885-020-07276-4. PMID 33028256
- [Derived] Noble SM, Garfield K, Lane JA, Metcalfe C, Davis M, Walsh EI, Martin RM, Turner EL, Peters TJ, Thorn JC, Mason M, Bollina P, Catto JWF, Doherty A, Gnanapragasam V, Hughes O, Kockelbergh R, Kynaston H, Paul A, Paez E, Rosario DJ, Rowe E, Oxley J, Staffurth J, Neal DE, Hamdy FC, Donovan JL. The ProtecT randomised trial cost-effectiveness analysis comparing active monitoring, surgery, or radiotherapy for prostate cancer. Br J Cancer. 2020 Sep;123(7):1063-1070. doi: 10.1038/s41416-020-0978-4. Epub 2020 Jul 16. PMID 32669672
- [Derived] Donovan JL, Opmeer B, Young GJ, Mills N, Martin RM, Lane JA, Metcalfe C, Peters TJ, Davis M, Turner EL, Walsh E, Neal DE, Hamdy FC; ProtecT Study Group. Factors associated with trial recruitment, preferences, and treatments received were elucidated in a comprehensive cohort study. J Clin Epidemiol. 2019 Sep;113:200-213. doi: 10.1016/j.jclinepi.2019.05.036. Epub 2019 Jun 3. PMID 31170515
- [Derived] Donovan JL, Young GJ, Walsh EI, Metcalfe C, Lane JA, Martin RM, Tazewell MK, Davis M, Peters TJ, Turner EL, Mills N, Khazragui H, Khera TK, Neal DE, Hamdy FC; ProtecT Study Group. A prospective cohort and extended comprehensive-cohort design provided insights about the generalizability of a pragmatic trial: the ProtecT prostate cancer trial. J Clin Epidemiol. 2018 Apr;96:35-46. doi: 10.1016/j.jclinepi.2017.12.019. Epub 2017 Dec 27. PMID 29288137
- [Derived] Young GJ, Harrison S, Turner EL, Walsh EI, Oliver SE, Ben-Shlomo Y, Evans S, Lane JA, Neal DE, Hamdy FC, Donovan JL, Martin RM, Metcalfe C. Prostate-specific antigen (PSA) testing of men in UK general practice: a 10-year longitudinal cohort study. BMJ Open. 2017 Oct 30;7(10):e017729. doi: 10.1136/bmjopen-2017-017729. PMID 29084797
- [Derived] Donovan JL, Hamdy FC, Lane JA, Mason M, Metcalfe C, Walsh E, Blazeby JM, Peters TJ, Holding P, Bonnington S, Lennon T, Bradshaw L, Cooper D, Herbert P, Howson J, Jones A, Lyons N, Salter E, Thompson P, Tidball S, Blaikie J, Gray C, Bollina P, Catto J, Doble A, Doherty A, Gillatt D, Kockelbergh R, Kynaston H, Paul A, Powell P, Prescott S, Rosario DJ, Rowe E, Davis M, Turner EL, Martin RM, Neal DE; ProtecT Study Group*. Patient-Reported Outcomes after Monitoring, Surgery, or Radiotherapy for Prostate Cancer. N Engl J Med. 2016 Oct 13;375(15):1425-1437. doi: 10.1056/NEJMoa1606221. Epub 2016 Sep 14. PMID 27626365
- [Derived] Hamdy FC, Donovan JL, Lane JA, Mason M, Metcalfe C, Holding P, Davis M, Peters TJ, Turner EL, Martin RM, Oxley J, Robinson M, Staffurth J, Walsh E, Bollina P, Catto J, Doble A, Doherty A, Gillatt D, Kockelbergh R, Kynaston H, Paul A, Powell P, Prescott S, Rosario DJ, Rowe E, Neal DE; ProtecT Study Group. 10-Year Outcomes after Monitoring, Surgery, or Radiotherapy for Localized Prostate Cancer. N Engl J Med. 2016 Oct 13;375(15):1415-1424. doi: 10.1056/NEJMoa1606220. Epub 2016 Sep 14. PMID 27626136
- [Derived] Wade J, Holding PN, Bonnington S, Rooshenas L, Lane JA, Salter CE, Tilling K, Speakman MJ, Brewster SF, Evans S, Neal DE, Hamdy FC, Donovan JL; ProtecT Study Group. Establishing nurse-led active surveillance for men with localised prostate cancer: development and formative evaluation of a model of care in the ProtecT trial. BMJ Open. 2015 Sep 18;5(9):e008953. doi: 10.1136/bmjopen-2015-008953. PMID 26384727
- [Derived] Kote-Jarai Z, Mikropoulos C, Leongamornlert DA, Dadaev T, Tymrakiewicz M, Saunders EJ, Jones M, Jugurnauth-Little S, Govindasami K, Guy M, Hamdy FC, Donovan JL, Neal DE, Lane JA, Dearnaley D, Wilkinson RA, Sawyer EJ, Morgan A, Antoniou AC, Eeles RA; UK Genetic Prostate Cancer Study Collaborators, and the ProtecT Study Group. Prevalence of the HOXB13 G84E germline mutation in British men and correlation with prostate cancer risk, tumour characteristics and clinical outcomes. Ann Oncol. 2015 Apr;26(4):756-761. doi: 10.1093/annonc/mdv004. Epub 2015 Jan 16. PMID 25595936
- [Derived] Oxley J, Simpkin A, Goepel J, Varma M, Griffiths D, Grigor K, Mayer N, Warren A, Deshmukh N, Bhattarai S, Dormer J, Hounsome L, Adamczyk LA, Metcalfe C, Lane JA, Davis M, Donovan JL, Neal DE, Hamdy FC, Robinson MC; ProtecT Study Group. Gleason drift in the NIHR ProtecT study. Histopathology. 2015 Feb;66(3):438-46. doi: 10.1111/his.12549. Epub 2015 Jan 7. PMID 25231130
- [Derived] Lane JA, Donovan JL, Davis M, Walsh E, Dedman D, Down L, Turner EL, Mason MD, Metcalfe C, Peters TJ, Martin RM, Neal DE, Hamdy FC; ProtecT study group. Active monitoring, radical prostatectomy, or radiotherapy for localised prostate cancer: study design and diagnostic and baseline results of the ProtecT randomised phase 3 trial. Lancet Oncol. 2014 Sep;15(10):1109-18. doi: 10.1016/S1470-2045(14)70361-4. Epub 2014 Aug 19. PMID 25163905
- [Derived] Fung-Kee-Fung SD, Porten SP, Meng MV, Kuettel M. The role of active surveillance in the management of prostate cancer. J Natl Compr Canc Netw. 2013 Feb 1;11(2):183-7. doi: 10.6004/jnccn.2013.0026. PMID 23411385
- See also: Project website — http://www.bristol.ac.uk/population-health-sciences/projects/protect/